CLINICAL TRIAL: NCT03660358
Title: Effect of Kinesiotaping Applications on Diaphragm, Abdomen and Chest Wall in Preterm Infants Undergoing Noninvasive Ventilation
Brief Title: Effect of Kinesiotaping Application in Preterm Infants Undergoing Noninvasive Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Associate Professor, Baskent University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA18/35
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Preterm Infant
Keywords: preterm infants; kinesiotape; ventilation; respiratory muscles
MeSH Terms: conditions — Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (Experimental): Kinesiotaping aplication to chest wall, abdomen and diaphragm in preterm infants.
  Interventions: Device: kinesiotape application
- Control (No Intervention): No kinesiotaping aplication to chest wall, abdomen and diaphragm in preterm infants.

INTERVENTIONS:
Device: kinesiotape application — kinesiotape application to diaphragm, chest wall and abdomen in preterm infants.
  Arms: Kinesiotape

SUMMARY:
Kinesiotaping (KT) applied to the thorax is believed to enhance breathing by supporting the respiratory muscles. Infants born premature usually have respiratory problems because of depletion of surfactant and respiratory muscle weakness. Therefore, we are going to use KT for premature infants in NICU who are undergoing non-invasive ventilation. Forty-two participants divided into two groups. The first group will be applied KT to chest wall, abdomen and diaphragm, and the other group will not receive any KT application during non-invasive ventilation. KT application will be going on as long as the infant underwent non-invasive ventilation. We are going to measure blood gas parameters (pH, pCO2, pO2, base excess), respiration rate, peak heart rate, percentage of Fio2, FiO2/pO2 rate, PEEP and PIP values before non-invasive ventilation, 2 hours after non-invasive ventilation, within 72 hours and shortly before weaning from non-invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient infants in NICU, born in Baskent University Ankara Hospital, undergoing non-invasive ventilation and age between 24-36.6 weeks.

Exclusion Criteria:

* Infants with multiple kongenital anomaly, hypoxic ischemic encephalopathy, tracheoesophageal fistula, diaphragmatic hernia.

Ages: 24 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
arterial blood gas | 1 day
  arterial blood gas

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ecevit, MD, Study Director — Associate Professor
Locations (1):
- Baskent University Ankara Hospital, Ankara, Bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No